CLINICAL TRIAL: NCT02525913
Title: Feasibility Study of Cavity Radiofrequency Ablation in ex Vivo Mastectomy Breast Tissue
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was withdrawn from the IRB and never opened. No subjects were enrolled.
Sponsor: University of Arkansas (Other)
Collaborators: Innoblative Designs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 204538
Record Dates: First submitted 2015-08-13; First posted 2015-08-18 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: Breast; Mastectomy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bi-lateral mastectomy (Other)
  Interventions: Device: RFA Applicator

INTERVENTIONS:
Device: RFA Applicator

SUMMARY:
The purpose of this study is to build a device that will consistently ablate (destroy or remove) cavitary breast tissue after a formal breast cancer resection in order to mimic the tissue that is now irradiated after breast cancer lumpectomy. The device would be easier to handle, perform the ablation in less time and by so ablating this margin would avoid the need in many for reoperation to obtain negative margins and based on preliminary data avoid the need for radiation. This would be especially important in poor and rural patients and would lead to decreased costs of treatment in patients with favorable breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age greater than or equal to 18 years.
* Receiving bi-lateral mastectomy due to tumor in the breast, or by choice (prophylactic mastectomy). Only non-cancerous breast tissue will be included in the study.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Those determined by the study investigator to have mental, physical, or medical conditions that would indicate that they should not participate.
* Because there is no patient contact with the device no medical contraindications are foreseen.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Ablation Depth | One year
  Ablation depth is the extent to which tissue has been completely desiccated from the wall of the cavity. It will be assessed by pathologic analysis using H&, PCNA, and Ki67 stains. The ablation depth of each slide processed is to be the smallest distance of completely necrotic tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Klimberg, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States